CLINICAL TRIAL: NCT02371291
Title: A Randomized Controlled Trial Comparing Memory Flexibility Training to Psychoeducation in the Treatment of Major Depressive Disorder
Brief Title: Memory Flexibility Training for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mrccbu
Record Dates: First submitted 2015-02-09; First posted 2015-02-25 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
Keywords: Memory Flexibility
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory Flexibility Training (Experimental): The MemFlex programme draws on cognitive bias modification and memory specificity training techniques (Raes et al., 2009; Dalgleish et al., 2014), and was developed by clinical psychologists. MemFlex is primarily self-guided and aims to reduce autobiographical memory biases associated with depression. The training material is presented over one face-to-face session and eight self-guided sessions. In the initial session, the researcher introduces cued-recall tasks which are used throughout the workbook, and guides the participant in completion of these tasks. When understanding of the basic principles is satisfactory, the researcher assists the participant to set a schedule for completion of the workbook over the following four weeks. The participant will receive weekly emails during this period, encouraging them to complete the workbook. They will also receive a phone call from a team member at the beginning of week three to check progress.
  Interventions: Behavioral: Memory Flexibility Training
- Psychoeducation (Placebo Comparator): The psychoeducation condition will also complete an initial face-to-face session. This session will cover the symptoms and causes of depression, and the workbook will be introduced. As in the MemFlex condition, the workbook will consist of eight self-guided sessions that the individual will be required to complete over four weeks. The participant will receive weekly emails during this period, encouraging them to complete the workbook. They will also receive a phone call from a team member at the beginning of week three to check progress, and clarify any difficulties with the workbook material. The workbook content will cover the presentation of depression and basic information on factors associated with depression, such as worry, procrastination, and sleep difficulties. Each session consists of information on psychological theories of the topic, followed by a series of questions about the material to ensure participant engagement. The workbook was developed by clinical psychologists.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Memory Flexibility Training — As in experimental arm description.
  Arms: Memory Flexibility Training
Behavioral: Psychoeducation — As in experimental arm description.
  Arms: Psychoeducation

SUMMARY:
Our collection of memories for personal experiences plays an important role in shaping our sense of who we are as people. These memories, termed autobiographical memories, can also be helpful in social situations, for sharing the details of our experiences with other people, reminiscing about pleasant times and solving problems by remembering what has and hasn't worked in the past. Different types of autobiographical memory are helpful to us depending on the particular situation the investigators are in at the time. Recent research has shown that experiencing depressed mood can affect how we relate to our autobiographical memories, so that instead of providing a rich source of personal information in a helpful and flexible way, the types of memories that come to mind are more narrowly focused on difficult or negative experiences. This can cause low mood to persist over time.

The purpose of this study is to test a newly-developed therapeutic training package for depressed mood (MemFlex), designed to encourage helpful and flexible ways of relating to autobiographical memories. The MemFlex programme consists of a one-to-one orientation session with the researcher to introduce the training package, followed by a workbook that is completed at home.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing Major Depressive Episode, indexed on the Structured Clinical Interview for the DSM-IV (SCID; First et al., 1996).
* Score of 13 or above on the Beck Depression Inventory (Beck et al., 1996)

Exclusion Criteria:

* SCID assessment indicates they are experiencing another mood disorder, psychosis, current alcohol or substance dependence/abuse.
* Diagnosed Axis II disorder or brain injury (assessed by participant report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Depressive Status | Three months after completion of the workbook
Change in score on the Beck Depression Inventory (Beck, Steer, & Brown, 1996) from baseline | Three months after completion of the workbook
  Self report measure of depression symptoms

SECONDARY OUTCOMES:
Depression free days | Three months after completion of the workbook
  Number of depression free days from post to follow-up.
Change in memory flexibility from baseline, Score on the alternating instructions autobiographical memory task (Dritschel et al., 2013) | Three months after completion of the workbook
  Score on the alternating instructions autobiographical memory task (Dritschel et al., 2013)

OTHER OUTCOMES:
Change in Rumination as measured by Rumination Response Scale | 4-6 weeks after beginning the workbook
  Rumination Response Scale (Treynor, Gonzalez, Nolen-Hoeksema, 2003);
Change in Cognitive Avoidance, as measured by Cognitive Avoidance Questionnaire | 4-6 weeks after beginning the workbook
  Cognitive Avoidance Questionnaire (Sexton & Dugas, 2008)
Change in Verbal Fluency as measured by the Verbal Fluency Task | 4-6 weeks after beginning the workbook
  Verbal Fluency Task
Change in Anxiety symptoms, as measured by the Beck Anxiety Inventory | 4-6 weeks after beginning the workbook
  Beck Anxiety Inventory
Change in Hopelessness, as measured by Beck Hopelessness Scale | 4-6 weeks after beginning the workbook
  Beck Hopelessness Scale
Change in Problem solving, as measured by the Means-Ends Problem Solving task | 4-6 weeks after beginning the workbook
  Means-Ends Problem Solving task (Lyubomirsky & Nolen-Hoeksema, 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dalgleish, PhD, Principal Investigator — MRC Cognition and Brain Sciences Unit
Locations (2):
- United Kingdom (2):
  - MRC Cognition and Brain Sciences Unit, Cambridge
  - Cambridge and Peterborough NHS Foundation Trust, Cambridge

REFERENCES:
- [Background] Raes F, Williams JM, Hermans D. Reducing cognitive vulnerability to depression: a preliminary investigation of MEmory Specificity Training (MEST) in inpatients with depressive symptomatology. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):24-38. doi: 10.1016/j.jbtep.2008.03.001. Epub 2008 Mar 12. PMID 18407245
- [Background] Dalgleish T, Bevan A, McKinnon A, Breakwell L, Mueller V, Chadwick I, Schweizer S, Hitchcock C, Watson P, Raes F, Jobson L, Werner-Seidler A. A comparison of MEmory Specificity Training (MEST) to education and support (ES) in the treatment of recurrent depression: study protocol for a cluster randomised controlled trial. Trials. 2014 Jul 22;15:293. doi: 10.1186/1745-6215-15-293. PMID 25052061
- [Background] Beck, A., Steer, R., & Brown, G. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] First, M., Spitzer, R., Gibbons, M., & Williams, J. (1996). Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-IV). Washington, DC: American Psychiatric Press.
- [Derived] Hitchcock C, Gormley S, Rees C, Rodrigues E, Gillard J, Panesar I, Wright IM, Hammond E, Watson P, Werner-Seidler A, Dalgleish T. A randomised controlled trial of memory flexibility training (MemFlex) to enhance memory flexibility and reduce depressive symptomatology in individuals with major depressive disorder. Behav Res Ther. 2018 Nov;110:22-30. doi: 10.1016/j.brat.2018.08.008. Epub 2018 Aug 29. PMID 30199738
- [Derived] Hitchcock C, Hammond E, Rees C, Panesar I, Watson P, Werner-Seidler A, Dalgleish T. Memory Flexibility training (MemFlex) to reduce depressive symptomatology in individuals with major depressive disorder: study protocol for a randomised controlled trial. Trials. 2015 Nov 3;16:494. doi: 10.1186/s13063-015-1029-y. PMID 26531124